CLINICAL TRIAL: NCT06576622
Title: Status Report on Periodontal Status and Oral Microbiota Women Who Have Suffered Repeated Miscarriages: a Pilot Study
Brief Title: PERIodontal Disease, Microbiota and Miscarriage
Acronym: PERI2M
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0053
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Miscarriage; Parodontitis
Keywords: REPEATED MISCARRIAGES; Porphyromonas gingivalis; SALIVA; BIOLOGICAL SAMPLES; subgingival plaque
MeSH Terms: conditions — Abortion, Spontaneous; Dry Socket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: biological sampling — As part of the health check-up oral, Will be taken:
  * Salivary samples by sputum.
  * Samples of subgingival plaque in the periodontal sulcus
  * A collection of the history and disease risk factors will then be carried out.
  * periodontal problems by a routine care interview, the clinical examination and radiological examination.

SUMMARY:
Cross-sectional non-interventional observational pilot study recruiting women whom had repeated miscarriages (= at least 3 miscarriages).The information will be collected during a routine maintenance, complete oral clinical and radiological examination (assessment carious, periodontal, mucosal and functional), which is part of the routine assessment in the service of odontology from Toulouse University Hospital.

Saliva and subgingival plaque samples, classically carried out in routine dental surgery as part of the health check-up oral, will be used to carry out bacterial assays.

DETAILED DESCRIPTION:
Cross-sectional non-interventional observational pilot study recruiting women whom had repeated miscarriages (= at least 3 miscarriages).The information will be collected during a routine maintenance, complete oral clinical and radiological examination (assessment carious, periodontal, mucosal and functional), which is part of the routine assessment in the service of odontology from Toulouse University Hospital.

As part of the health check-up oral, Will be taken:

* Salivary samples by sputum (1 per patient). The patient will retain her saliva for 1 minute in the mouth and it will be collected in a sterile bottle (approximately 5 ml).
* Samples of subgingival plaque in the periodontal sulcus (assessed during periodontal probing) using sterile paper points (minimum 3 and maximum 10 per patient) inserted for 30 seconds into the periodontal sulcus then put in a tube sterile. The plate collection is done by capillary action on the paper tip, a very small quantity is thus taken.

A collection of the history and disease risk factors will then be carried out. periodontal problems (stress level assessed using the visual analogue scale, history personal and family periodontal diseases, oral hygiene habits, etc.) by a routine care interview, the clinical examination (visual examination and recording of oral and periodontal) and radiological examination.

ELIGIBILITY:
Inclusion Criteria:

* women whom had repeated miscarriages
* at least 6 natural teeth

Exclusion Criteria:

* under antibiotic prebiotic or probiotics treatment one month prior to the study
* with high infection risk (HIV,...)

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women whom had repeated miscarriages
Study Population: women whom had repeated miscarriages : at least 3
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
average quantity of Porphyromonas gingivalis | AT INCLUSION = T0
  estimate the average quantity of Porphyromonas gingivalis (Pg) in saliva patients who have had recurrent miscarriages (3 consecutive miscarriages < 14 weeks of amenorrhea)

SECONDARY OUTCOMES:
microbiological composition | AT INCLUSION = T0
  microbiological composition of the saliva in women having had repeated miscarriages :
  Salivary samples by sputum (1 per patient). The patient will retain her saliva for 1 minute in the mouth and it will be collected in a sterile bottle (approximately 5 ml).
microbiological composition | AT INCLUSION = T0
  microbiological composition of the subgingival plaque in women having had repeated miscarriages
  Samples of subgingival plaque in the periodontal sulcus (assessed during periodontal probing) using sterile paper points (minimum 3 and maximum 10 per patient) inserted for 30 seconds into the periodontal sulcus then put in a tube sterile. The plate collection is done by capillary action on the paper tip, a very small quantity is thus taken.

CONTACTS AND LOCATIONS:
Locations (1):
- UH Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No